CLINICAL TRIAL: NCT01840943
Title: A Phase 3, Randomized, Open-Label, Comparative Bridging Study of CAELYX® Versus Topotecan HCl in Subjects With Epithelial Ovarian Carcinoma Following Failure of First-Line, Platinum-Based Chemotherapy
Brief Title: A Study to Compare CAELYX With Topotecan HCL in Patients With Recurrent Epithelial Ovarian Carcinoma Following Failure of First-Line, Platinum-Based Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the study was terminated due to medication supply issue from current manufacturer
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100654; DOXILOVC3001 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2013-03-18; First posted 2013-04-26 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial ovarian cancer; Recurrent epithelial ovarian carcinoma; Carcinoma; Malignancy; Ovarian carcinoma; CAELYX; Topotecan hydrochloride; Topotecan; Platinum-based regimen chemotherapy; Chinese patients
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Carcinoma; Neoplasms; Ovarian Neoplasms | interventions — liposomal doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAELYX (Experimental): Participants will receive CAELYX 50 mg per square meter intravenously on Day 1 of each cycle as: 60 to 90-minute infusion to the participants not undergoing pharmacokinetic (PK) evaluation and 90-minute infusion to the participants undergoing PK evaluation.
  Interventions: Drug: CAELYX
- Topotecan hydrochloride (HCl) (Active Comparator): Participants will receive topotecan HCl 1.25 mg per square meter per day, intravenously for 30-minutes duration, on Day 1 to Day 5 of each cycle.
  Interventions: Drug: Topotecan HCl

INTERVENTIONS:
Drug: CAELYX — CAELYX 50 mg per square meter will be administered intravenously on Day 1 of each cycle as: 60 to 90-minute infusion to the participants not undergoing pharmacokinetic (PK) evaluation and 90-minute infusion to the participants undergoing for PK evaluation.
  Arms: CAELYX
Drug: Topotecan HCl — Topotecan 1.25 mg per square meter per day will be administered, intravenously for 30-minutes duration, on Day 1 to Day 5 of each cycle.
  Arms: Topotecan hydrochloride (HCl)

SUMMARY:
The purpose of this study is to compare the effectiveness between CAELYX and topotecan hydrochloride (HCl) in Chinese participants with recurrent epithelial ovarian carcinoma following failure of first-line, platinum-based chemotherapy, who have received no more than one prior platinum-based regimen therapy.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), comparative bridging study (a supplemental study which performs to provide data of effectiveness, safety, and dosage to compare two study medications in a new region). The study consists of 3 phases: screening phase (30 days before administration of study medication), treatment phase, and follow up phase (every 8 weeks for tumor assessment until disease progression or death, or until the study completion, whichever is earlier and every 3 months after disease progression for overall survival and for anti-tumor therapy for a minimum of 1 year). In the treatment phase, approximately 120 eligible participants will be categorized prospectively for platinum-sensitivity (sensitive versus refractory) and bulky disease (presence versus absence). Later on participants will be randomly assigned either to experimental arm (CAELYX: administer on Day 1 of each cycle) or control arm (topotecan HCl: administer on Day 1 to Day 5 of each cycle). Treatment will continue until disease progression occurs and may continue for at least 2 cycles after confirmed complete response (disappearance of all target lesions). On average, it is expected that participants will continue treatment for approximately 3 to 6 cycles in experimental arm (CAELYX) or 4 to 8 cycles in Control arm (topotecan HCl). Safety evaluations will include assessment of adverse events, clinical laboratory tests, electrocardiogram, echocardiogram (or multiple gated acquisition scans), vital signs, and physical examination which will be monitored throughout the study. The total duration of the study will be approximately 23 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosed with epithelial ovarian carcinoma with measurable disease
* Recurrent epithelial ovarian carcinoma or disease progression following failure of first-line, platinum-based chemotherapy with no more than one prior platinum based regimen therapy
* Adequate laboratory values of bone marrow function, renal function, liver function, and echocardiogram tests
* Agrees to use protocol-defined effective contraception. A woman must agree not to donate eggs (ova, oocytes) for the purpose of assisted reproduction
* Disease-free from prior malignancies for more than 5 years with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix

Exclusion Criteria:

* Females who are pregnant or breast feeding or planning to become pregnant while enrolled in this study or within 1 year after the last dose of study medication
* Myocardial infarct within 6 months before enrollment, class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
* Uncontrolled systemic infection that requires systemic anti-infective treatment
* Prior therapy with CAELYX or topotecan HCl
* Prior chemotherapy within 28 days of first dose of study medication (or 42 days if participant has received a nitrosourea or mitomycin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (7):
- China (7):
  - Beijing
  - Changsha
  - Guangzhou
  - Jinan
  - Nanjing
  - Nanning
  - Wuhan

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 32 participants screened, 26 were randomized to study treatment.
Groups:
- CAELYX: Participants received 50 milligram per square meters (mg/m^2) of Caelyx as a 90-minute or 60 to 90-minute intravenous infusion every 4 weeks.
- Topotecan Hydrocloride (HCl): Participants received topotecan HCl 1.25 mg per square meter per day, intravenously for 30-minutes duration, on Day 1 to Day 5 of each cycle.
Period: Overall Study
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Started | 14 | 12
Completed | 1 | 0
Not Completed | 13 | 12
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Physician Decision | 4 | 2
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat population included (mITT) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl) | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (4.97) | 51.6 (8.32) | 54.0 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival Incidence at Week 24
Description: Progression-free survival incidence was be measured as number of participants who were progression-free and alive. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20 percent (%) increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Week 24
Population: The modified intent-to-treat population included (mITT) included all randomized participants.
Measure: Number; unit: participants
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 14 | 12
participants | 6 | 2

2. Secondary Outcome: Duration of Progression-free Survival
Description: It was calculated as the time, in weeks, from the day of randomization until documented disease progression or death due to any cause, whichever occurs first using a Kaplan-Meier curve for PFS.
Time Frame: 1 year after the last dose (24 weeks) administration
Population: The mITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 14 | 12
weeks | NA [8.0 to NA] — Insufficient number of participants with events. | 24.6 [7.9 to 25.1]

3. Secondary Outcome: Number of Participants With Response
Description: Response rate was measured as number of participants with at least a durable response: Complete response (CR) or partial response (PR). Complete response is defined as the disappearance of all target lesions. Partial response is defined as at least a 30 percentage decrease in the sum of diameters of target lesions. Stable disease defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Progression in disease is defined as at least a 20% increase in the sum of diameters of target lesions. Not evaluable participants were those who were not analyzed. The reference of the baseline sum of diameters of lesions was considered.
Time Frame: Up to Week 24
Population: The mITT population included all randomized participants.
Measure: Number; unit: participants
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 14 | 12
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 5 | 3
  Stable Disease (SD) | 4 | 6
  Progression Disease (PD) | 1 | 1
  Not Evaluable (NE) | 4 | 2

4. Secondary Outcome: Time to Response
Description: It is calculated as the day of randomization to the first observation of a durable response (the first of the 2 confirmatory measurements).
Time Frame: Up to Week 24
Population: The mITT population included all randomized participants.Time to response was analyzed for participants who achieved response.
Measure: Median (Full Range); unit: weeks
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 5 | 3
weeks | 16.0 [8.0 to 24.1] | 16.0 [6.0 to 16.1]

5. Secondary Outcome: Duration of Response
Description: It is calculated as the first observation of a durable response (the first of the 2 confirmatory measurements) to the first observation of disease progression or death due to any cause.
Time Frame: Up to 1 year of last dose (Week 24) administration
Population: The mITT population included all randomized participants. Duration of response was analyzed for participants who achieved response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 5 | 3
weeks | NA [8.1 to NA] — Insufficient number of participants with events. | 9.3 [8.6 to 10.6]

6. Secondary Outcome: Health-related Quality of Life Assessment (HQL)
Description: Calculation of each HQL domain scale will be performed according to the scoring guidelines for each of the HQL measures. The HQL analyses will include scales measuring physical functioning, pain, nausea, fatigue, and global quality of life. Each item is measured on a scale of 0 to 3, where 0 = no impact on quality of life and 3 = extreme impact on quality of life.
Time Frame: Day 1 of each cycle of study medication and Week 4 after last dose of study medication
Population: Data was not collected for this outcome measure as the study was early terminated.
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Overall Survival
Description: Number of Participants With Overall survival were categorized as number of 1) Deaths, 2) Still alive, 3) Early termination from the study due to lost to follow up, 4) Early termination from the study due to withdraw of consent, 5) Other. Overall survival is defined as the time interval from randomization to death from any cause.
Time Frame: Week 4 after the last dose of the study medication and approximately up to 1 year after the disease progression or completion of the study treatment or death, whichever is earlier
Population: The mITT population included all randomized participants.
Measure: Number; unit: participants
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 14 | 12
participants
  Death | 1 | 0
  Still alive | 0 | 0
  Early termination: due to lost to follow up | 4 | 4
  Early termination: due to withdraw of consent | 5 | 6
  Other | 4 | 2

8. Secondary Outcome: Maximum Plasma Concentration of CAELYX
Time Frame: 0 hour, 30 minutes, 90 minutes, 2 hours, 4 hours, 8 hours, 12 hours, Day 2, Day 3, Day 5, Day 8, and Day 11 for Cycle 1 and Cycle 2
Population: Data was not collected for this outcome measure as the study was early terminated.
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Reach the Maximum Plasma Concentration of CAELYX
Time Frame: as for outcome 8
Population: Data was not collected for this outcome measure as the study was early terminated.
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Area Under the Plasma Concentration of CAELYX
Time Frame: as for outcome 8
Population: Data was not collected for this outcome measure as the study was early terminated.
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Apparent Terminal Elimination Half-life of Plasma Concentration of CAELYX
Time Frame: as for outcome 8
Population: Data was not collected for this outcome measure as the study was early terminated.
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Apparent Terminal Elimination Rate Constant of Plasma Concentration of CAELYX
Time Frame: as for outcome 8
Population: Data was not collected for this outcome measure as the study was early terminated.
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Systemic Clearance of Plasma Concentration of CAELYX
Time Frame: as for outcome 8
Population: Data was not collected for this outcome measure as the study was early terminated.
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Apparent Volume of Distribution of Plasma Concentration of CAELYX
Time Frame: as for outcome 8
Population: Data was not collected for this outcome measure as the study was early terminated.
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Grade 3 (Severe) events are symptoms causing inability to perform usual social & functional activities. Grade 4 (Life-threatening) events are Symptoms causing inability to perform basic self-care functions or Medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death.
Time Frame: Up to 30 days after the last dose of study medication
Population: Safety population included all randomized participants.
Measure: Number; unit: participants
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Number analyzed (Participants) | 14 | 12
participants
  TEAEs | 12 | 12
  TESAEs | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study medication
Description: Safety population included all randomized participants.
Arm/Group | CAELYX | Topotecan Hydrocloride (HCl)
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/12
Other Adverse Events (participants affected / at risk) | 12/14 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAELYX (N=14) | Topotecan Hydrocloride (HCl) (N=12)
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAELYX (N=14) | Topotecan Hydrocloride (HCl) (N=12)
Anemia (Blood and lymphatic system disorders) | 5 | 11
Leukopenia (Blood and lymphatic system disorders) | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Leukocytosis (Investigations) | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
White blood cell count decreased (Investigations) | 6 | 10
Neutrophil count decreased (Investigations) | 6 | 9
Platelet count decreased (Investigations) | 0 | 6
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Weight decreased (Investigations) | 1 | 1
Blood albumin decreased (Investigations) | 1 | 0
Lymphocyte percentage decreased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 8
Nausea (Gastrointestinal disorders) | 6 | 5
Constipation (Gastrointestinal disorders) | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Folliculitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Infusion related reaction (Immune system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early as the total number of participants treated in this study was low and only descriptive analysis was used for efficacy and safety evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.